CLINICAL TRIAL: NCT05389241
Title: Monocentric Prospective Randomized Study on the Influence of On-screen Use of a Virtual 3-dimensional Liver Model Reconstructed From CT Data on Spatial Perception During Laparoscopy on the Liver Phantom.
Brief Title: Laparoscopic Augmented Reality for Identification of Liver Lesions - a Pre-clinical Randomized Cross-over Trial
Acronym: LARA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Principal Investigator, Roger Wahba, MD, PhD, Priv.-Doz. Dr. med Roger Wahba, Universitätsklinikum Köln
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 21-1406
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Laparoscopy; Augmented Reality; Orientation, Spatial; Liver
Keywords: Augmented reality; liver; minimally invasive surgery; laparoscopy; 3D; spatial orientation; digital health; artificial intelligence
MeSH Terms: conditions — Orientation, Spatial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Method A (Experimental): Subjects in this arm will perform the task on the liver phantom with Method A (2D-CT). Then they will do the NASA task load index questionnaire. After that they will perform the tasks with Method B (2D-CT + 3D augmented reality model). After that again a NASA Task load index questionnaire is performed
  Interventions: Other: Method A
- Method B (Experimental): Subjects in this arm will perform the task on the liver phantom with method B (2D-CT + 3D augmented reality model). Then they will do the NASA task load index questionnaire. After that they will perform the tasks with Method A (2D-CT). After that again a NASA Task load index questionnaire is performed
  Interventions: Other: Method B

INTERVENTIONS:
Other: Method A — The subjects will perform tasks on the liver phantom (identification of target lesions). They will perform the tasks with Method A (2D-CT) or Method B (2D-CT + 3D augmented reality model). the intervention type Method A means that the trainings set up is performed first with Method A an after that with Method B.
  Arms: Method A
Other: Method B — The subjects will perform tasks on the liver phantom (identifikation of target lesions). They will perform the tasks with Method A (2D-CT) or Method B (2D-CT + 3D augmented reality model). the intervention type Method B means that the trainings set up is performed first with Method B an after that with Method A.
  Arms: Method B

SUMMARY:
Procedure preparation and accurate knowledge of the specific anatomy is an integral part of performing minimally invasive procedures. Due to the complexity with high variability and the non-visibility of the vascular structures, the liver poses a particular challenge.

Therefore medical students and experienced surgeons will receive standardized, structured training on liver anatomy, the use of laparoscopic ultrasound and the application and use of CT data sets and the virtual 3D liver model. This training will be evaluated by questionnaires. Both groups then carry out a series of localization exercises on an artificial liver phantom: tumor imitations, which are displayed in the image(3D virtaul mdoel or 2D-CT-Data-Set), have to be found in the liver phantom laparoscopically using ultrasound.

In each round, different scenarios are worked on, once without and then with the support of the virtual 3D liver model. The virtual 3D model can be displayed directly on the laparoscopic monitor using a display software specially developed for the trial and can be manipulated by the subjects.

The aim of the study is to provide evidence that the availability and use of a virtual 3D model (augmented reality) leads to a significantly improved spatial perception of the subjects during laparoscopy of the liver. In addition, the subjectively perceived cognitive load of the subjects during the test run with and without the support of the virtual 3D model is surveyed and the learning success is evaluated.

DETAILED DESCRIPTION:
Procedure preparation and accurate knowledge of the specific anatomy is an integral part of performing a minimally invasive procedure. Due to the complexity with high variability and the non-visibility of the vascular structures due to the location in the parenchyma, the liver poses a particular challenge. The spatial perception and cognitive processing of the anatomical target structures is of particular importance.

The aim of this study is to test the hypothesis that the use of a 3-dimensional (3D) virtual liver model (virtual 3D model crating augmented reality) presenedt on teh laparoscopic screeen reconstructed from CT data exerts an influence on the spatial perception of subjects during laparoscopy on the liver phantom.

After informed consent and consent to the study, a pseudonymised subject population consisting of surgeons with experience in laparoscopy (n=36) and an equal number of medical students without experience in laparoscopy (n=36) will be included in the study included. The subjects will be randomized and divided into two groups of equal size, stratified according to experience in laparoscopy. The randomization is carried out by a data trustee. All subjects then receive standardized, structured training on liver anatomy, the use of laparoscopic ultrasound, and the application and use of CT data sets and the virtual 3D liver model. This is evaluated by means of a questionnaire. Both groups then sequentially carry out a defined series of localization exercises on an artificial liver phantom: tumor imitations, which are displayed in the image, have to be found in the liver phantom laparoscopically using ultrasound. In each round, different scenarios are worked on once without and then with the support of the virtual 3D liver model. The virtual 3D model can be displayed directly on the laparoscopic monitor using display software specially made for the study and can be manipulated by the subjects. The aim of the study is to provide evidence that the availability and use of a virtual 3D model leads to a significantly improved spatial perception of the subjects during laparoscopy of the liver. In addition, the subjectively perceived cognitive load of the subjects during the test run with and without the support of the virtual 3D model is surveyed by NASA Task Load Index and the learning success is evaluated.

The primary endpoints of the study are the number of correctly spatially identified target structures and the time required to localize the given target structures.

ELIGIBILITY:
Inclusion Criteria:

* medical student of University of Cologne OR medical doctor in a surgical specialty
* informed consent signed

Exclusion Criteria:

* known and not correctable deficit of stereoscopic view
* for medical students: experience with laparoscopy or laparoscopy simulators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of correctly identified targets | immediately after tasks are performed, Day 1
  The number of correctly spatially identified targets (tumors in the liver phantom)
Time required | immediately after tasks are performed, Day 1
  The time required to localize the specified target structures (tumors in the live phantom)

SECONDARY OUTCOMES:
Task Load Index | immediately after tasks are performed, Day 1
  The specific cognitive effort of the subject (measured using the NASA Task Load Index)
Modification of procedure planning | immediately after tasks are performed with both methods, Day 1
  The modification of the initially prepared procedure planning when the virtual 3D model is available
Learning curve | immediately after tasks are performed with both methods, Day 1
  Qualitative evaluation of the learning curve and success of the subjects

CONTACTS AND LOCATIONS:
Overall Officials: Roger Wahba, MD, PHD, Principal Investigator — Universitätsklinikum Köln
Locations (1):
- University of Cologne, Department of General, Visceral and Cancer Surgery, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No